CLINICAL TRIAL: NCT07131163
Title: Neoadjuvant Chemo-immunotherapy Not Resected
Brief Title: Real World Stage II-III NSCLC Patients Receiving Neoadjuvant Chemo-immunotherapy and no Surgical Resection
Acronym: NoSurgery
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other); Soroka University Medical Center (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Hadassah Medical Organization (Other); Rabin Medical Center (Other); University Hospital, Geneva (Other); Tel-Aviv Sourasky Medical Center (Other Government); MedStar Georgetown University Hospital (Other); Mayo Clinic (Other); UOMi Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2172-25-SMC; 8993-11-SMC (Other: Sheba Medical Center)
Record Dates: First submitted 2025-08-03; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Stage II-III Non-small Cell Lung Cancer
Keywords: neoadjuvant; NSCLC; Non-small-cell lung cancer; immunotherapy; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients who started neoadjuvant chemo-immontherapy followed by cancellation of surgery: Stage II-III NSCLC patients who started neoadjuvant chemo-immontherapy between January 1st 2022 to September 30th 2024 followed by cancellation of surgery

SUMMARY:
Neoadjuvant chemo-immunotherapy, with or without adjuvant immunotherapy, is currently the standard of care for resectable stage II-III NSCLC. One of the major drawbacks of neoadjuvant treatment is the risk of surgery cancellation. In most of the studies including a neoadjuvant component of treatment, about 20% of recruited patients do not undergo surgery. The reasons for surgery cancellation are recorded as a mixture of adverse events, disease progression, patient's decision and physician's decision. There is lack of data about the precise reasons for cancellation of the surgery. For patients starting neoadjuvant chemo-immunotherapy followed be cancellation of surgery, there is lack of data about the need to add additional treatments and about outcome of these treatments. Depending on the reason for surgery cancellation, these patients might undergo salvage radiotherapy (or chemo-radiotherapy), switch to systemic treatment as for metastatic disease or to palliative care.

Goal of the study: to collect real-world data about NSCLC patients that started neoadjuvant chemo-immunotherapy and did not get to surgery.

Study conduct Participating centers will secure approvals for retrospective collection of clinical data. Relevant patients will be identified from the working database of each center, data will be collected locally, deidentified and collected centrally at the Sheba MC.

Data collected will include: demographics (age, sex); patients' characteristics (smoking status, co-morbidities, ECOG-PS, weight loss); tumor characteristics (histology, molecular tests, specific test results, clinical stage); staging procedures done (CT, PET-CT, brain MRI, EBUS, mediastinoscopy); neoadjuvant treatment (regimen, number of cycles, dose reductions, delays); reason for surgery cancellation; to be categorized according to the following options: iRAE/ non-immune-related AEs/ molecular test results/ re-staging result showing lack of mediastinal clearing/ distant disease progression/ local progression leading to patient becoming not-resectable/ re-assessment of patient as not-resectable (without a significant change in the tumor)/ change in the patient condition making the patient not-operable.

Major Inclusion criteria:

1. Stage II-III NSCLC patient, based on clinical staging.
2. Treated by a chemo-immunotherapy regimen defined as neoadjuvant treatment, for at least one cycle of treatment.
3. No surgery was performed for at least six months from initiation of the neoadjuvant treatment.

DETAILED DESCRIPTION:
1. Participating centers will secure an ethics and administrative approval for retrospective collection of clinical data.
2. Relevant patients will be identified from the working database of each center, data will be collected locally, deidentified and collected centrally.
3. Where required, patients will be requested to provide informed consent for the participation in the study.
4. Data collected will include

   1. Demographics (age, sex)
   2. Patients' characteristics (smoking status, co-morbidities, ECOG-PS, weight loss)
   3. Tumor characteristics (histology, molecular tests, specific test results, clinical stage).
   4. Staging procedures done (CT, PET-CT, brain MRI, EBUS, mediastinoscopy)
   5. Neoadjuvant treatment (regimen, number of cycles, dose reductions, delays).
   6. Reason for surgery cancellation; to be categorized according to the following options:

   i. iRAE, ii. non-immune-related AEs, iii. molecular test result, iv. re-staging result showing lack of mediastinal clearing, v. distant disease progression, vi. local progression leading to patient becoming not-resectable, vii. re-assessment of patient as not-resectable (without a significant change in the tumor), viii. change in the patient condition making the patient not-operable.
5. Data will be entered to an eCRF, anonymized and collected centrally at Sheba MC.
6. Analysis of the data according to the statistical analysis plan.

Inclusion criteria:

1. Stage II-III NSCLC patient, based on clinical staging.
2. Treated by a chemo-immunotherapy regimen defined as neoadjuvant treatment, for at least one cycle of treatment.
3. No surgery was performed for at least six months from initiation of the neoadjuvant treatment.
4. Availability of data about reasons for surgery cancellation and clinical follow up.
5. Patient's consent for data collection (or waiver of the need for consent by the local ethics committee).
6. At least 6 mo of follow up after initiation of neoadjuvant treatment.

Statistical analysis plan:

Data will be analyzed based on the reason defined for surgery cancellation. Analyses will be descriptive, reporting mean, median, 95% C.I. as relevant. Time-to-event measures will be estimated by Kaplan-Meier method. Comparisons between groups will be done in a descriptive manner, using t-test, Chi-square and log-rank test as appropriate.

Ethics: Each participating center will receive approval of the local IRB. Unless waived, each participating patient will sign an informed consent form prior to any study procedure.

Patient data confidentiality: No identifying information regarding participating patients will leave each of the centers. Participants will be given a study code, the key connecting the code to the patients' identity will be kept at each participating site secured as per local regulations of each site.

Data transfer: clinical data files (excel or equivalent) will be transferred to Sheba MC by email.

Data sharing: At the end of the study, the clinical data will be made available to requesting researchers following review of requests.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II-III NSCLC patient, based on clinical staging.
2. Treated by a chemo-immunotherapy regimen defined as neoadjuvant treatment, for at least one cycle of treatment.
3. No surgery was performed for at least six months from initiation of the neoadjuvant treatment.
4. availability of data about reasons for surgery cancellation and clinical follow up.
5. patient's consent for data collection (or waiver of the need for consent by the local ethics committee)
6. At least 6 month of follow up after intiation of neoadjuvant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage II-III NSCLC patient who have started neoadjuvant chemo-immunotherapy between January 1st 2022 to September 30th 2024.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of patients that do not undergo surgery after initiating NACT-IO | Up to 6 months after initation of NACT-IO
  Percentage of patients who do not reach surgery after initiating NACT-IO
Causes for surgery cancellation | Up to 6 months after initation of NACT-IO
  Percentage of patients whose surgery is cancelled regarding: Toxicity, disease progression, unresectable, inoperable, other causes.

CONTACTS AND LOCATIONS:
Overall Officials: Jair Bar, MD-PhD, Principal Investigator — Jusidman Cancer Center, Sheba Medical Center
Locations (1):
- Jusidman Cancer Center, Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Based on direct communication with study officials
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting from study publication for 2 years.
Access Criteria: Based on direct communication with study officials